CLINICAL TRIAL: NCT06671379
Title: A Randomized, Open-label, Multicenter, Phase III Study of SHR-A2009 Versus Platinum-based Chemotherapy in EGFR-mutated, Advanced or Metastatic Non-small Cell Lung Cancer After Failure of Epidermal Growth Factor Receptor (EGFR) Tyrosine Kinase Inhibitor (TKI) Therapy
Brief Title: A Study of SHR-A2009 Versus Platinum-based Chemotherapy in EGFR-mutated, Advanced or Metastatic NSCLC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A2009-301
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A2009 monotherapy (Experimental)
  Interventions: Drug: SHR-A2009 monotherapy
- platinum-based dual-agent chemotherapy (Active Comparator)
  Interventions: Drug: platinum-based dual-agent chemotherapy

INTERVENTIONS:
Drug: SHR-A2009 monotherapy — SHR-A2009 monotherapy ，SHR-A2009 will be administered intravenously
  Arms: SHR-A2009 monotherapy
Drug: platinum-based dual-agent chemotherapy — Pemetrexed combined with carboplatin or cisplatin, after four cycles of combination, pemetrexed was continued as a single agent，all drugs will be administered intravenously
  Arms: platinum-based dual-agent chemotherapy

SUMMARY:
This study was a randomized, controlled, open-label, multicenter phase III clinical study to compare the efficacy and safety of SHR-A2009 with platinum-based dual-agent chemotherapy in patients with EGFR-mutated advanced or metastatic non-small cell lung cancer who failed EGFR TKI treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old (inclusive), Female or male
2. Subjects with unresectable locally advanced or metastatic non-squamous non-small cell lung cancer confirmed by histology or cytology
3. Previously treated by EGFR-TKI；
4. At least one measurable tumor lesion according to RECIST v1.1
5. ECOG performance score of 0-1;
6. Expected survival time ≥ 12 weeks;
7. Adequate bone marrow and organ function
8. Subjects are required to give informed consent for this study prior to the trial and voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Subjects with active central nervous system (CNS) metastases.
2. Received antitumor therapy such as chemotherapy within 4 weeks prior to the first dose of study drug;
3. Received >30 Gy of non-thoracic radical radiation therapy within 4 weeks prior to the first administration of study drug;
4. Major organ surgery or significant trauma within 4 weeks prior to first use of study drug;
5. Concomitant other malignancies ≤ 5 years prior to first dose of study drug;
6. Subjects with a history of interstitial pneumonitis or imaging at screening suggestive of suspected interstitial pneumonitis; or other moderate-to-severe lung disease that severely affects lung function
7. Serious cardiovascular disease
8. Presence of severe infection within 4 weeks prior to first dose of study drug
9. Arterial/venous thrombotic events within 3 months prior to the first study dose
10. History of immunodeficiency, including a positive HIV test
11. Presence of active hepatitis B or C;
12. History of allergic reactions to any component of study treatment or severe allergic reactions to other monoclonal antibodies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by BICR according to RECIST v1.1 | Up to approximately 32 months

SECONDARY OUTCOMES:
overall survival (OS) | Up to approximately 32 months
Progression Free Survival(PFS by investigator) | Up to approximately 32 months
Duration of response(DoR，by BICR and investigator ) | Up to approximately 32 months
Disease control rate（DCR，by BICR and investigator） | Up to approximately 32 months
Incidence of AEs | from Day1 to 40 days after last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided